CLINICAL TRIAL: NCT02092766
Title: Parenteral Artesunate Compared to Quinine as a Cause of Late Post-treatment Anaemia in African Children With Hyperparasitaemic P. Falciparum Malaria
Brief Title: Parenteral Artesunate Compared to Quinine as a Cause of Late Anaemia in African Children With Malaria
Acronym: DHART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Kinshasa School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KIMORU005
Record Dates: First submitted 2014-03-13; First posted 2014-03-20 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Anaemia
Keywords: malaria; anaemia; artesunate
MeSH Terms: conditions — Anemia; Malaria | interventions — Artesunate; Quinine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV artesunate (Experimental): Intravenous artesunate 2.4 mg/kg body weight STAT, then 2.4 mg/kg at 12, 24, 48 and 72 hours (5 doses total)
  Interventions: Drug: artesunate
- IV quinine (Active Comparator): Intravenous quinine dihydrochloride 20 mg salt/kg body weight loading dose over 4 hours, then 10 mg/kg over 2 hours 8 hourly until 72 hours (9 doses total)
  Interventions: Drug: quinine

INTERVENTIONS:
Drug: artesunate
  Arms: IV artesunate
Drug: quinine
  Arms: IV quinine

SUMMARY:
Delayed anaemia has been reported in European travellers with malaria cured by artesunate. Although no deaths related to this delayed anaemia have been reported so far, blood transfusion has been necessary in some affected patients. Recent observations suggest that this episodes of anaemia also occurs in endemic countries. The aim of this trial is to assess the incidence of late onset anaemia after treatment with intravenous artesunate compared to intravenous quinine, to identify patients at risk and to clarify the causes of this delayed anaemia.

ELIGIBILITY:
Inclusion Criteria:

* Age > 6 months and ≤ 14 years
* Acute uncomplicated P. falciparum malaria, confirmed by positive blood smear with asexual forms of P. falciparum or mixed with non-falciparum species
* Asexual P. falciparum parasitaemia ≥ 100,000/uL and ≤500,000/uL
* Haemoglobin ≥5.0 g/dL
* Parents/guardians agree to hospitalize the child for the length of treatment (3 days) and bring the patient for planned follow-up visits at day 7, 14, 21, 28, 35, 42
* Signed consent from the guardian/parents

Exclusion Criteria:

* Body weight ≤ 5 kg
* Severe malaria or signs of severe malaria as defined by WHO Guidelines 2013
* History of hypersensitivity or contraindication to quinine or artesunate
* A clear history of adequate antimalarial treatment in the preceding 24 hours with drugs expected to be effective
* Presence of intercurrent illness or any condition which in the judgement of the investigator would place the subject at undue risk or interfere with the patient treatment or results of the study
* Participation in another clinical trial

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 217 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Late onset anaemia | Patients are hospitalized for 4 days or longer if still unwell. After discharge the follow-up consists of 6 weekly visits (time frame 42 days). Late anaemia is measured between 7 and 42 days following the start of antimalarial treatment
  Late onset anaemia in this study is defined as a ≥10% drop in haemoglobin on any previous measurement anytime between day 7 and 42

CONTACTS AND LOCATIONS:
Locations (1):
- Kinshasa School of Public Health, Kinshasa, Democratic Republic of the Congo

REFERENCES:
- [Derived] Fanello C, Onyamboko M, Lee SJ, Woodrow C, Setaphan S, Chotivanich K, Buffet P, Jaureguiberry S, Rockett K, Stepniewska K, Day NPJ, White NJ, Dondorp AM. Post-treatment haemolysis in African children with hyperparasitaemic falciparum malaria; a randomized comparison of artesunate and quinine. BMC Infect Dis. 2017 Aug 17;17(1):575. doi: 10.1186/s12879-017-2678-0. PMID 28818049